CLINICAL TRIAL: NCT06524401
Title: Novel Post-Surgical Incision Management to Prevent Ostomy Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A22-066
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Ostomy; Enterocutaneous Fistula
Keywords: Stoma; Ileostomy
MeSH Terms: conditions — Intestinal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Limpet (Experimental): Participants in this arm will utilize the subject device as intended to be used.
  Interventions: Device: Limpet
- Control (Active Comparator): Standard treatment with standard of care adhesive ostomy pouches.
  Interventions: Device: Control

INTERVENTIONS:
Device: Limpet — Limpet participants will have their device placed by a clinician. Upon discharge, a portable vacuum pump will be issued to provide negative pressure (e.g., 3M Prevena or Snap; ConvaTec Avelle; or Pensar MicroDoc). These systems are compact, fit in a pocket, are simple to operate, and commonly used in the outpatient setting to provide multiple weeks of therapy. Participants will be furnished with materials to address potential dressing problems while at home: extra waste pouches, adhesive drape strips for sealing air leaks, and standard of care adhesive ostomy pouches and accessories as a backup plan in the event of a Limpet failure.
  Arms: Limpet
Device: Control — Control participants will receive standard of care adhesive ostomy pouch dressings. Participants will be furnished with materials to address potential dressing problems while at home: adhesive ostomy pouches and accessories for pouch replacement. The Control group will change their pouches at home 2 to 5 times per week or more frequently if needed, as per the current standard of care.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of the Limpet, as compared to standard of care ostomy pouches, in reducing complications for ostomy and fistula patients. Secondary objectives include evaluating dressing leak rates and causes of complications (e.g., edema, tissue oxygen saturation, and poor stoma eversion). The main questions it aims to answer are:

Primary Hypothesis 1: Peristomal Skin Complications will decrease

Primary Hypothesis 2: Dressing Leak Rates will decrease

Participants will:

* Receive either the Limpet device or standard of care adhesive ostomy pouch dressing
* Return every 7 days for study visits for 30 days to receive device replacement, wound imaging, blood tests, and quality of life surveys.

DETAILED DESCRIPTION:
The Limpet is a single-use device intended for effluent management and promotion of healing of intact and injured skin surrounding enterocutaneous fistulae and ostomies.

Our study focuses on small bowel openings, encompassing two important cohorts: 1) ileostomy and 2) enterocutaneous fistulas (ECFs). Our study's success criterion is primarily based on the pooled results from both cohorts.

Primary Hypothesis 1: Peristomal Skin Complications (PSCs): We hypothesize that the Limpet will demonstrate a significant improvement in PSCs compared to standard of care adhesive ostomy pouches. Specifically, we anticipate a raw difference of 35% in PSCs for the pooled cohorts, with a complication rate of 50% in the control group and 15% in the Limpet group.

Primary Hypothesis 2: Dressing Leak Rates: We hypothesize that the Limpet will demonstrate a significant improvement in dressing leak rates compared to standard of care adhesive ostomy pouches. Specifically, we anticipate a raw difference of 15% in leak rates for the pooled cohorts, with a leak rate of 30% in the control group and 15% in the Limpet group.

These hypotheses are grounded in existing literature, supplemented by clinical experience. We intend to conduct subgroup analyses to assess the treatment effect across the two cohorts (ileostomy and ECF) and across other relevant subgroups such as gender, race, etc.

Secondary Hypothesis: Total Complications (PSCs and Stomal Complications): We hypothesize that the Limpet will exhibit a raw difference of 35% in total complications (comprising PSCs and stomal complications like mucocutaneous separation and stoma retraction) for the ileostomy cohort. Stoma complication rates vary widely in the literature, and we plan to conduct sub analyses to evaluate the Limpet's effect on stoma complications independent of PSCs.

This will be a 30 day, single-site, randomized controlled trial (RCT) for a non-significant risk device, Limpet.

The study will have a two-arm parallel group design:

* Limpet: Participants in this arm will utilize the subject device as intended to be used.
* Control: Standard treatment with standard of care adhesive ostomy pouches.

Ninety-two participants (78 stoma and 14 enterocutaneous fistula participants) will be randomized after they have consented to study participation. Initial randomization will occur in a 1:1 ratio (Limpet and Control). Participants will be randomly stratified with permuted blocks by BMI (≤ vs > 40) and stoma type (loop ileostomy, end ileostomy, or enterocutaneous fistula) to account differences in healing and wound severity.

This study will be conducted at HealthPartners Institute's Regions Hospital in St. Paul, Minnesota. Data compiled by the Wound, Ostomy, and Continence Nursing Department reveals an annual pool of more than 300 eligible patients at Regions Hospital.

The study will consist of the following visits:

* Visit C1 (Day -35 to -6): Screening in-person clinic visit
* Visit C2, Day 1: Baseline appointment clinic visit
* Visit C3, Week 1: Clinic visit
* Visit C4, Week 2: Clinic visit
* Visit C5, Week 3: Clinic visit
* Visit C6, Week 4: Final appointment during treatment period; clinic visit

After the Baseline Data Collection Period, participants will be randomized by BMI and three stoma types: ileostomy with loop stoma, ileostomy with end stoma, and enterocutaneous fistulas (ECFs) into 1 of 2 treatment groups:

* Limpet: Participants in this arm will utilize the subject device as intended to be used.
* Control: Standard treatment with standard of care adhesive ostomy pouches.

On Day 1, Limpet participants will have their device placed by a clinician. Upon discharge, a portable vacuum pump will be issued to provide negative pressure (e.g., 3M Prevena or Snap; ConvaTec Avelle; or Pensar MicroDoc). These systems are compact, fit in a pocket, are simple to operate, and commonly used in the outpatient setting to provide multiple weeks of therapy. Participants will be furnished with materials to address potential dressing problems while at home: extra waste pouches, adhesive drape strips for sealing air leaks, and standard of care adhesive ostomy pouches and accessories as a backup plan in the event of a Limpet failure.

On Day 1, Control participants will receive standard of care adhesive ostomy pouch dressings. Participants will be furnished with materials to address potential dressing problems while at home: adhesive ostomy pouches and accessories for pouch replacement. The Control group will change their pouches at home 2 to 5 times per week or more frequently if needed, as per the current standard of care.

The brand and model of pumps and adhesive ostomy pouches used by Limpet and Control participants will be recorded for comparison purposes. Participants will return for clinic visits approximately every 7 days to have their device replaced. Participants will have their final study appointment approximately 30 days post-surgery. Clinical support will help the participant troubleshoot dressing problems; and if necessary, bring the patient into the study site for an immediate dressing change.

ELIGIBILITY:
Inclusion Criteria:

* Participant is greater than 18 years of age, inclusive
* Participant is undergoing ileostomy surgery or,
* has an enterocutaneous fistula with output over 500cc in 24 hours
* Participants stoma will have a maximum diameter of 1.5 inches based on measurements from the Investigator or Sponsor.
* Area around the stoma must have no injury through the dermis (i.e., intact skin)
* Participant is willing and able to comply with all protocol-specified requirements
* Participant is capable of reading and understanding English and will provide written informed consent to participate.

Exclusion Criteria:

* Unable/unwilling to attend the follow-up appointments
* Participant has a life expectancy < 30 days.
* Participant has a stature too small for use of the Limpet in the opinion of the Investigator or Sponsor.
* Participant has an enteroatmospheric fistula (enteric fistula to an open wound)
* Participant is scheduling/planning concurrent chemotherapy or other radiation treatment during the study follow-up period
* Participant has a history of sensitivity or allergy to hydrocolloids or other materials in the Limpet device.
* Participant is pregnant or planning to become pregnant (verbal report).
* Participant is unable or unwilling to provide informed consent.
* Participant is currently participating in an investigational drug or another device study that clinically interferes with the current study endpoints.
* Participant has any other disease or medical condition that, in the opinion of the Investigator or Sponsor, could endanger the participant, interfere with the evaluation of the study device's efficacy or safety, or compromise the participant's ability to comply with/complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Peristomal Skin Complications (PSCs) | 30 days
  We hypothesize that the Limpet will demonstrate a significant improvement in PSCs compared to standard of care adhesive ostomy pouches. Specifically, we anticipate a raw difference of 35% in PSCs for the pooled cohorts, with a complication rate of 50% in the control group and 15% in the Limpet group.
Dressing Leak Rates | 30 Days
  We hypothesize that the Limpet will demonstrate a significant improvement in dressing leak rates compared to standard of care adhesive ostomy pouches. Specifically, we anticipate a raw difference of 15% in leak rates for the pooled cohorts, with a leak rate of 30% in the control group and 15% in the Limpet group.

SECONDARY OUTCOMES:
Total Complications (PSCs and Stomal Complications) | 30 Days
  We hypothesize that the Limpet will exhibit a raw difference of 35% in total complications (comprising PSCs and stomal complications like mucocutaneous separation and stoma retraction) for the ileostomy cohort. Stoma complication rates vary widely in the literature, and we plan to conduct sub analyses to evaluate the Limpet's effect on stoma complications independent of PSCs.

CONTACTS AND LOCATIONS:
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with external entities outside of aggregate form for publication. Deidentified data will be shared with the study sponsor. Study identifiers will be destroyed after publication.